CLINICAL TRIAL: NCT00615459
Title: A Phase III, Randomized, Double-blind, Double-dummy, Placebo-controlled, Multicenter, 3-period Incomplete Block, Multidose Crossover Study to Determine the Effect on Lung Function of Indacaterol (150 and 300 μg o.d.) in Patients With Moderate to Severe COPD, Using Tiotropium (18 μg o.d.) as an Active Control
Brief Title: A Crossover Study to Determine the Effect on Lung Function of Indacaterol in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD), Using Tiotropium as an Active Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CQAB149B2331
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic obstructive pulmonary disease, indacaterol, tiotropium, placebo controlled
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1: Placebo,Tiotropium, Indacaterol 150 μg (Experimental): In period I, placebo to indacaterol (150 or 300 μg) delivered via SDDPI. The placebo for blinding tiotropium was delivered via the tiotropium inhalation device. In period II, tiotropium (18 μg) once daily delivered via inhalation device and matching placebo to indacaterol delivered once daily via single dose dry powder inhaler (SDDPI). In period III, indacaterol 150 μg once daily delivered via SDDPI and placebo to tiotropium was delivered once daily via the tiotropium inhalation device. Daily inhaled corticosteroid (ICS) monotherapy (where applicable) was provided to remain stable throughout study. The Short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Tiotropium; Drug: Placebo
- Sequence 2: Indacaterol 300 μg, Indacaterol 150 μg, Tiotropium (Experimental): In period I,indacaterol 300 μg once daily delivered via single dose dry powder inhaler (SDDPI)and matching placebo to tiotropium delivered once daily via tiotropium inhalation device. In period II, indacaterol 150 μg once daily delivered via SDDPI and matching placebo to tiotropium delivered once daily via tiotropium inhalation device. In period III, tiotropium (18 μg) once daily delivered via inhalation device and matching placebo to indacaterol delivered once daily via SDDPI. Daily ICS monotherapy (where applicable) was provided to remain stable throughout study. The SABA was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Tiotropium
- Sequence 3: Indacaterol 150 μg, Indacaterol 300 μg, Placebo (Experimental): In period I, indacaterol 150 μg once daily delivered via SDDPI and matching placebo to tiotropium delivered once daily via tiotropium inhalation device. In period II, indacaterol 300 μg once daily delivered via SDDPI and matching placebo to tiotropium delivered once daily via tiotropium inhalation device. In period III, placebo to indacaterol (150 or 300 μg) delivered via SDDPI. The placebo for blinding tiotropium was delivered via the tiotropium inhalation device. Daily ICS monotherapy (where applicable) was provided to remain stable throughout study. The SABA was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Placebo
- Sequence 4: Tiotropium, Placebo, Indacaterol 300 μg (Experimental): In period I, tiotropium (18 μg) once daily delivered via inhalation device and matching placebo to indacaterol delivered once daily via SDDPI. In period II, placebo to indacaterol (150 or 300 μg) delivered via SDDPI. The placebo for blinding tiotropium was delivered via the tiotropium inhalation device. In period III, indacaterol 300 μg once daily delivered via SDDPI and matching placebo to tiotropium delivered once daily via tiotropium inhalation device. Daily ICS monotherapy (where applicable) was provided to remain stable throughout study. The SABA was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Tiotropium; Drug: Placebo

INTERVENTIONS:
Drug: Indacaterol — Indacaterol 150 μg or 300 μg, delivered via SDDPI
Drug: Tiotropium — Tiotropium 18 μg once daily delivered via inhalation device
  Arms: Sequence 1: Placebo,Tiotropium, Indacaterol 150 μg; Sequence 2: Indacaterol 300 μg, Indacaterol 150 μg, Tiotropium; Sequence 4: Tiotropium, Placebo, Indacaterol 300 μg
Drug: Placebo — Placebo to indacaterol (150 or 300 μg) delivered via SDDPI. The placebo for blinding tiotropium was delivered via the tiotropium manufacturer's proprietary inhalation device (HandiHaler®)
  Arms: Sequence 1: Placebo,Tiotropium, Indacaterol 150 μg; Sequence 3: Indacaterol 150 μg, Indacaterol 300 μg, Placebo; Sequence 4: Tiotropium, Placebo, Indacaterol 300 μg

SUMMARY:
The study compared the 24-hour spirometry profile of indacaterol with that of placebo and with tiotropium as an active control in patients with chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged ≥ 40 years, who have signed an Informed Consent Form prior to initiation of any study-related procedure
* Co-operative out patients with a diagnosis of chronic obstructive pulmonary disease (COPD) (moderate to severe as classified by the Global initiative for chronic obstructive lung disease (GOLD) Guidelines, 2006) and:

  1. Smoking history of at least 10 pack years (current or previous smokers)
  2. Post-bronchodilator forced expiratory volume in 1 second (FEV1) < 80% and ≥30% of the predicted normal value.
  3. Post-bronchodilator FEV1/Forced vital capacity (FVC) < 70%

Exclusion Criteria:

* Patients who have been hospitalized for a COPD exacerbation in the 6 weeks prior to Visit 1 or during the run-in period
* Patients requiring long-term oxygen therapy for chronic hypoxemia
* Patients who have had a respiratory tract infection within 6 weeks prior to Visit
* Patients with concomitant pulmonary disease
* Patients with a history of asthma
* Patients with diabetes Type I or uncontrolled diabetes Type II
* Any patient with lung cancer or a history of lung cancer
* Any patient with active cancer or a history of cancer with less than 5 years disease free survival time
* Patients with a history of long QT syndrome or whose QTc interval (Bazett's) measured at Visit 1 or randomization is prolonged
* Patients who have been vaccinated with live attenuated vaccines within 30 days prior to screening or during the run-in period.
* Patients unable to successfully use a dry powder inhaler device, MDI or perform spirometry measurements

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma, Study Chair — Novartis Pharmaceuticals
Locations (20):
- Novartis Investigative site, Camperdown, Australia
- Germany (5):
  - Novartis Investigator Site, Gauting
  - Novartis Investigator Site, Großhansdorf
  - Novartis Investigator Site, Mainz
  - Novartis Investigator site, Marburg
  - Novartis Investigator Site, Wiesbaden
- Netherlands (5):
  - Novartis Investigator Site, Almelo
  - Novartis Investigator Site, Breda
  - Novartis Investigator Site, Eindhoven
  - Novartis Investigator Site, Harderwijk
  - Novartis Investigator Site, Helmond
- Novartis Investigator Site, Wellington, New Zealand
- Poland (2):
  - Novartis Investigator Site, Katowice
  - Novartis Investigator Site, Warsaw
- Novartis Investigator Site, Durban, South Africa
- Spain (5):
  - Novartis Investigator Site, A Coruña
  - Novartis Investigative site, Alicante
  - Novartis Investigative Site, Cacenes
  - Novartis Investigative Site, Madrid
  - Novartis Investigator Site, Ourense

REFERENCES:
- [Derived] Vogelmeier C, Ramos-Barbon D, Jack D, Piggott S, Owen R, Higgins M, Kramer B; INTIME study investigators (INdacaterol & TIotropium: Measuring Efficacy). Indacaterol provides 24-hour bronchodilation in COPD: a placebo-controlled blinded comparison with tiotropium. Respir Res. 2010 Oct 5;11(1):135. doi: 10.1186/1465-9921-11-135. PMID 20920365

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized to one of the 4 possible treatment sequences of the double-blind 10-week treatment phase (Week 1 - 10) to receive three out of the four study treatments. Each treatment sequence was divided into three 2-week treatment periods (I/II/III), with periods I and II followed by 2-week washout periods.
Pre-assignment Details: Out of total 169 randomized patients, two patients were discontinued before exposure to any treatment in period I because of administrative problems.
Period: Period I
Arm/Group | Sequence 1: Placebo,Tiotropium, Indacaterol 150 μg | Sequence 2: Indacaterol 300 μg, Indacaterol 150 μg, Tiotropium | Sequence 3: Indacaterol 150 μg, Indacaterol 300 μg, Placebo | Sequence 4: Tiotropium, Placebo, Indacaterol 300 μg
Started | 41 | 41 (1 randomized patient of this sequence was never exposed to drug. Hence, dropped out before Period I.) | 42 (1 randomized patient of this sequence was never exposed to drug. Hence, dropped out before Period I.) | 43
Completed | 37 | 40 | 40 | 42
Not Completed | 4 | 1 | 2 | 1
Not completed — Adverse Event | 2 | 0 | 1 | 0
Not completed — Subject withdrew consent | 1 | 0 | 0 | 1
Not completed — Abnormal test procedure results | 1 | 1 | 1 | 0
Period: Period II
Arm/Group | Sequence 1: Placebo,Tiotropium, Indacaterol 150 μg | Sequence 2: Indacaterol 300 μg, Indacaterol 150 μg, Tiotropium | Sequence 3: Indacaterol 150 μg, Indacaterol 300 μg, Placebo | Sequence 4: Tiotropium, Placebo, Indacaterol 300 μg
Started | 37 | 40 | 40 | 42
Completed | 36 | 40 | 40 | 41
Not Completed | 1 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Period: Period III
Arm/Group | Sequence 1: Placebo,Tiotropium, Indacaterol 150 μg | Sequence 2: Indacaterol 300 μg, Indacaterol 150 μg, Tiotropium | Sequence 3: Indacaterol 150 μg, Indacaterol 300 μg, Placebo | Sequence 4: Tiotropium, Placebo, Indacaterol 300 μg
Started | 36 | 40 | 40 | 41
Completed | 36 | 37 | 39 | 41
Not Completed | 0 | 3 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Administrative problems | 0 | 1 | 1 | 0
Not completed — Unsatisfactory therapeutic effect | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Patients: The safety population, included all patients who received at least one dose of study drug.
Arm/Group | Total Patients
Number analyzed (Participants) | 167
Age Continuous [Mean (Standard Deviation); unit: years] | 64.5 (7.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 128

OUTCOME MEASURES:

1. Primary Outcome: 24-hour Post-dose Trough Forced Expiratory Volume in 1 Second (FEV1) After 14 Days of Treatment
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. Trough FEV1 was defined as the mean of FEV1 measurements at 23 h 10 min and 23 h 45 min post Day 14 dose measured on the morning of Day 15 in each treatment period. The model used for analysis contained the (period) baseline FEV1 as covariate. The (period) baseline FEV1 was defined as the value measured before the study drug administration in that treatment period.
Time Frame: 23 hours 10 minutes and 23 hours 45 minutes post-dose on Day 15 of each treatment period
Population: The modified intent-to-treat (mITT) population, included all randomized patients who received at least one dose of study drug. Patients were analyzed according to treatment they received.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Indacaterol 150 μg: Indacaterol 150 μg once daily delivered via SDDPI and placebo to tiotropium was delivered once daily via the tiotropium inhalation device. Daily inhaled corticosteroid (ICS) monotherapy (where applicable) was provided to remain stable throughout study. The Short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
- Indacaterol 300 μg: Indacaterol 300 μg once daily delivered via single dose dry powder inhaler (SDDPI)and matching placebo to tiotropium delivered once daily via tiotropium inhalation device. Daily inhaled corticosteroid (ICS) monotherapy (where applicable) was provided to remain stable throughout study. The Short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
- Tiotropium 18 μg: Tiotropium (18 μg) once daily delivered via inhalation device and matching placebo to indacaterol delivered once daily via single dose dry powder inhaler (SDDPI). Daily inhaled corticosteroid (ICS) monotherapy (where applicable) was provided to remain stable throughout study. The Short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
- Placebo: Placebo to indacaterol (150 or 300 μg) delivered via SDDPI. The placebo for blinding tiotropium was delivered via the tiotropium inhalation device. Daily inhaled corticosteroid (ICS) monotherapy (where applicable) was provided to remain stable throughout study. The Short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
Arm/Group | Indacaterol 150 μg | Indacaterol 300 μg | Tiotropium 18 μg | Placebo
Number analyzed (Participants) | 116 | 119 | 112 | 118
Liters | 1.53 (0.021) | 1.51 (0.021) | 1.48 (0.021) | 1.36 (0.021)

2. Secondary Outcome: Peak FEV1 During 4 Hours Post Morning Dose on Day 1
Description: FEV1 was measured with spirometry conducted according to internationally accepted standards. The peak effect on Day 1 was defined as the maximum FEV1 during the first 4 hour on that day. FEV1 measurements taken within 6 hour of rescue use were set to missing before the peak FEV1 (0-4 hour) was calculated. The model used for analysis contained the (period) baseline FEV1 as covariate. The (period) baseline FEV1 was defined as the value measured before the study drug administration in that treatment period.
Time Frame: Day 1 (from 0 to 4 hours post morning dose)
Population: The modified intent-to-treat (mITT) population, included all randomized patients who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol 150 μg | Indacaterol 300 μg | Tiotropium 18 μg | Placebo
Number analyzed (Participants) | 118 | 122 | 120 | 121
Liters | 1.65 (0.015) | 1.67 (0.015) | 1.62 (0.015) | 1.48 (0.015)

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: In the safety population, all patients were analyzed according to treatment received.
Groups:
- Indacaterol 150 μg: Indacaterol 150 μg once daily delivered via single dose dry powder inhaler (SDDPI) and placebo to tiotropium was delivered once daily via the tiotropium inhalation device. Daily inhaled corticosteroid (ICS) monotherapy (where applicable) was provided to remain stable throughout study. The short acting (beta) β2-agonist (SABA) was available for rescue use throughout the study.
- Indacaterol 300 μg: Indacaterol 300 μg once daily delivered via single dose dry powder inhaler (SDDPI). Daily ICS monotherapy (where applicable) was provided to remain stable throughout study. The SABA was available for rescue use throughout the study.
- Tiotropium 18 μg: Tiotropium 18 μg once daily delivered via inhalation device. Daily ICS monotherapy (where applicable) was provided to remain stable throughout study. The SABA was available for rescue use throughout the study.
- Placebo: Placebo to indacaterol (150 or 300 μg) delivered via SDDPI. The placebo for blinding tiotropium was delivered via the tiotropium inhalation device. Daily ICS monotherapy (where applicable) was provided to remain stable throughout study. The SABA was available for rescue use throughout the study.
Arm/Group | Indacaterol 150 μg | Indacaterol 300 μg | Tiotropium 18 μg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/118 | 1/122 | 4/120 | 1/123
Other Adverse Events (participants affected / at risk) | 15/118 | 17/122 | 11/120 | 13/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 μg (N=118) | Indacaterol 300 μg (N=122) | Tiotropium 18 μg (N=120) | Placebo (N=123)
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol 150 μg (N=118) | Indacaterol 300 μg (N=122) | Tiotropium 18 μg (N=120) | Placebo (N=123)
Nasopharyngitis (Infections and infestations) | 4 | 9 | 5 | 6
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 7 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.